CLINICAL TRIAL: NCT06916962
Title: Understanding Psycho-socioeconomic Linkages Through an Intervention Providing Enhanced Financial and Social Support During Tuberculosis Treatment
Brief Title: Examining Psycho-Socioeconomic Linkages in TB Care: The UPLIFT Trial
Acronym: UPLIFT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Freundeskreis Für Internationale Tuberkulosehilfe e.V (Other)
Collaborators: Karolinska Institutet (Other); Liverpool School of Tropical Medicine (Other); Vietnam National Lung Hospital (Unknown); Korea International Cooperation Agency (KOICA) (Unknown); Stop TB (Unknown)
Responsible Party: Principal Investigator, Rachel Forse, Program Director, Freundeskreis Für Internationale Tuberkulosehilfe e.V
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21/25/CN-HDDD-BVPTU
Record Dates: First submitted 2025-03-12; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Tuberculosis (TB)
Keywords: Low- and Middle-income Countries; Treatment support; Catastrophic costs; Psychosocial support; Cash transfers; Health-related quality of life; Social protection
MeSH Terms: conditions — Tuberculosis | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Participants will be individually randomized using a non-blinded stratified randomization approach to allocate sub-groups of participants (by gender and recruitment site) into the intervention or control group, in a 1:1 ratio.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Participants in this arm will receive standard care TB treatment delivered by Vietnam's National TB Program (NTP), which includes routine counseling, support, and materials. Highly vulnerable individuals will be eligible to access existing government financial assistance through established mechanisms and eligibility criteria. No cash transfers will be received by control group participants, nor will they be invited to participate in TB Clubs.
- Intervention (Experimental): Intervention participants will receive the psycho-socioeconomic intervention.
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Intervention — Intervention participants will receive cash transfers on the condition of their participation in peer-led TB support meetings (TB Clubs).
  Two monthly TB Club meetings will be held in each participating district. Each will aim to provide enhanced education about the TB treatment process, as well as to improve treatment engagement and adherence, foster social support and mitigate TB-related stigma.
  Participants will be eligible for a maximum of three cash transfers, amounting to a total of 3,000,000 VND. The first payment of 1,000,000 VND will be made after a participant joins one TB Club, the second payment will be completed after attending a second TB Club, and the third payment will be provided after attendance at their 6th TB Club.
  Other Names: Psycho-socioeconomic support
  Arms: Intervention

SUMMARY:
Introduction: Tuberculosis (TB) remains an ongoing public health and socioeconomic challenge worldwide, especially in low- and middle-income countries such as Vietnam. Despite improvements in healthcare, TB still causes significant problems to those infected, especially within marginalized populations, including financial hardship, stigma, and mental health issues. This study aims to assess the effectiveness of a psycho-socioeconomic support intervention intended to improve treatment outcomes and reduce financial hardship faced by TB-affected households in Vietnam, measured through catastrophic costs.

Methods: A hybrid type II effectiveness implementation study using a randomized control trial study design will be employed to evaluate the effectiveness and implementation of the intervention. The study will be conducted in 12 Vietnamese provinces across Northern, Central, and Southern regions, targeting areas with lower TB treatment success rates. Participants will be randomly assigned to either a control group, which will receive standard care, or an intervention group, which will receive cash transfers conditioned on participation in TB Club peer-support meetings. Data will be collected on the individual, household and district levels. Individual outcomes will include treatment success, health-related quality of life, TB-related stigma, and anxiety and depression. Household outcomes will include catastrophic cost incurrence, changes in financial capital and livelihoods, and TB service and universal health coverage (UHC) uptake. Implementation outcomes, by district, will include fidelity, satisfaction, participation, acceptability, and quality.

Hypothesis: The study hypothesizes that providing financial and enhanced psychosocial support to people with TB will improve their treatment success and reduce the financial burden on TB-affected households.

DETAILED DESCRIPTION:
Background - Previous Studies on Social Protection for TB in Vietnam

This study has been designed based on the results of previous formative research on the preferences, acceptability, and feasibility of TB-specific social protection interventions in the Vietnamese context. This body of research found that people with TB and healthcare providers prefer cash transfers and enrollment in Vietnam's social health insurance scheme, especially when targeted to those with the greatest financial need and severe illness. A pilot study was conducted that provided cash transfers and social health insurance to economically vulnerable people starting TB treatment. The intervention was found broadly acceptable, but stakeholders felt that cash-transfers should be subject to limited forms of conditionality. Findings from this pilot indicated that future socioeconomic interventions in Vietnam should consider both conditional and unconditional cash transfers to be feasible.

Following this pilot, a non-randomized social assistance intervention was conducted under programmatic conditions. Among the group receiving financial support, it was found that a combination of transport vouchers, cash transfers and health insurance enrollment, combined with existing government and social network support could reduce catastrophic costs by 37.8%.

Finally, a one-year consultative process was conducted in 2023 to co-prioritize challenges and solutions with Vietnam's TB Program. This process found that an intervention supplementing the existing social safety net with TB-specific support was the priority.

Methods - Sample Size Two sample sizes were calculated to determine the effectiveness of the intervention. The larger sample will be used to recruit individuals undergoing TB treatment to measure changes in TB treatment success, while a subset of these same individuals will be recruited to assess catastrophic cost incurrence in the household, which will utilize a modified, longitudinal WHO TB Patient Cost Survey tool. A total of 1,324 participants (662 per study arm) will be recruited for the treatment success sample, while 450 (225 per study arm) will be recruited for the household costing sample.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with drug-sensitive, pulmonary, new, or relapse TB
* Initiated on TB treatment and reported/notified in VITIMES
* Residing in one of the implementation districts for the past 1 month
* First member of the household to enroll in the study

Exclusion Criteria:

* Not enrolled in VITIMES within 1 month of treatment initiation
* Household registration in another province
* Plans to relocate in the next 6 months
* Additional family members living in the same household with someone enrolled in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1324 (Estimated)
Dates: Start 2025-03-14 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
TB Treatment Success | Through study completion, an average of 6 months.
  Difference in the proportion of those cured or completing treatment between the two study arms
Catastrophic costs | The period from the onset of TB symptoms through study completion, an average of 9 months.
  Difference in the proportion of households where the combined direct and indirect costs of TB treatment-after accounting for any financial support received-amount to ≥20% of their estimated pre-treatment household income.
Composite fidelity score | 1 year
  Level of adherence to the design of the intervention components (cash transfers conditioned on TB Club participation) including the content, coverage, frequency, and duration, by district. The composite fidelity score has been structured according to Carroll et al. (2007) A conceptual framework for implementation fidelity.

SECONDARY OUTCOMES:
Health-Related Quality of Life | Through study completion, an average of 6 months.
  Difference in the health-related quality of life of study participants between the two arms, as measured by EuroQoL's EQ-5D-5L.
TB-Related Stigma | Through study completion, an average of 6 months.
  Difference in the perceived TB-related stigma reported by participants between the two study arms, as measured by the Redwood scale for TB-related stigma in Vietnam.
Financial Capital | The period from the onset of TB symptoms through study completion, an average of 9 months.
  Changes in financial capital such as dissavings, asset sales, borrowing and social support, between the two study arms. The definition of financial capital will be taken from Timire et al. (2023) Use of a Sustainable Livelihood Framework-Based Measure to Estimate Socioeconomic Impact of Tuberculosis on Households.
Sustainable Livelihood | The period from the onset of TB symptoms through study completion, an average of 9 months.
  Difference in livelihood impacts such as food insecurity and educational disruptions, between the two study arms. The definition of this outcome will be taken from Timire et al. (2023) Use of a Sustainable Livelihood Framework-Based Measure to Estimate Socioeconomic Impact of Tuberculosis on Households.
TB Service and UHC Uptake | Through study completion, an average of 6 months.
  Difference in the proportion of household members screened for TB, initiating preventive therapies or purchasing social health insurance, between the two study arms.
Implementation quality score | 1 year
  During two-week time windows, implementation districts will be scored with up to 5 points for implementation quality, and quality scores for each window and district will be averaged to obtain an intervention quality score by district, province and region. Quality will be defined as timeliness of intervention delivery and participant satisfaction with the intervention at each district.
Participation | 1 year
  Average number of TB Clubs attended per participant, within each district.
Acceptability | 1 year
  Acceptability of the intervention as measured by district. Acceptability will be defined by Sekhon et al. (2022) Development of a theory-informed questionnaire to assess the acceptability of healthcare interventions.

CONTACTS AND LOCATIONS:
Locations (12):
- Vietnam (12):
  - Long Dien District TB Unit, Ba Ria Vung Tau
  - O Mon District TB Unit, Can Tho
  - Lien Chieu District TB Unit, Da Nang
  - Son Tra District TB Unit, Da Nang
  - Phuc Tho District TB Unit, Hanoi
  - Binh Chanh District TB Unit, Ho Chi Minh City
  - District 04 District TB Unit, Ho Chi Minh City
  - District 5 District TB Unit, Ho Chi Minh City
  - Hoc Mon District TB Unit, Ho Chi Minh City
  - Can Duoc District TB Unit, Long An
  - Tan Hung District TB Unit, Long An
  - Thang Binh District TB Unit, Điện Bàn

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Forse R, Yoshino CA, Nguyen TT, Phan THY, Vo LNQ, Codlin AJ, Nguyen L, Hoang C, Basu L, Pham M, Nguyen HB, Van Dinh L, Caws M, Wingfield T, Lonnroth K, Sidney-Annerstedt K. Towards universal health coverage in Vietnam: a mixed-method case study of enrolling people with tuberculosis into social health insurance. Health Res Policy Syst. 2024 Apr 2;22(1):40. doi: 10.1186/s12961-024-01132-8. PMID 38566224
- [Background] Forse R, Nguyen TT, Dam T, Vo LNQ, Codlin AJ, Caws M, Minh HDT, Nguyen LH, Nguyen HB, Nguyen NV, Lonnroth K, Annerstedt KS. A qualitative assessment on the acceptability of providing cash transfers and social health insurance for tuberculosis-affected families in Ho Chi Minh City, Vietnam. PLOS Glob Public Health. 2023 Dec 6;3(12):e0002439. doi: 10.1371/journal.pgph.0002439. eCollection 2023. PMID 38055709
- [Background] Smith I, Forse R, Sidney Annerstedt K, Thanh NT, Nguyen L, Phan THY, Nguyen H, Codlin A, Vo LNQ, Nguyen NTT, Khan A, Creswell J, Pham Huy M, Basu L, Lonnroth K, Nguyen BH, Nguyen VN, Atkins S. What matters most? A qualitative study exploring priorities for supportive interventions for people with tuberculosis in urban Viet Nam. BMJ Open. 2023 Aug 23;13(8):e076076. doi: 10.1136/bmjopen-2023-076076. PMID 37612116
- See also: Related Info — https://tbhelp.org